CLINICAL TRIAL: NCT01322217
Title: Network-Wide Assessment of Current Health Status and Behavioral Risk Factors: An Expanded Study for New Sites in ATN III
Brief Title: Managerial Database II
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: ATN 106
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-03

CONDITIONS: Acquired Immunodeficiency Syndrome
Keywords: Medication adherence; Substance use; Sexual risk behaviors
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AMTU Clients: All HIV-infected adolescents and young adults engaged in care at sites newly participating in ATN III and their affiliates who are between 12 and 24 years of age, inclusive, are aware of their HIV status and understand written and/or verbal English will be eligible for inclusion in the study. In addition, new patients who have their initial clinic visit within the enrollment period will also be eligible for participation.

SUMMARY:
This study will collect information on health status and risk behaviors, as well as basic demographic and biomedical information for a group of HIV positive adolescents receiving care at sites newly participating in ATN III.

DETAILED DESCRIPTION:
The proposed study is a cross sectional study intended to be conducted at each of the Adolescent Medicine Trials Units (AMTUs) newly participating in ATN III and to enroll all participating patients followed at each site. This approach will allow for the examination of the broad spectrum of youth participating in the ATN, including those newly entered into care.

Psychosocial and risk-taking behavioral data will be collected using Audio Computer-Assisted Self-Interview (ACASI) for English-speaking participants, or a paper-and-pencil Spanish-language survey with identical measures to the ACASI for Spanish-speaking participants; biomedical information will be collected through medical chart abstraction.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory evidence of HIV-1 infection documented by a positive result on any of the following licensed tests at any time: Any HIV-1 antibody test confirmed by Western blot, HIV-1 culture, HIV-1 DNA PCR, or plasma HIV-1 RNA PCR > 1,000 copies/ml;
* Knowledge of HIV positive diagnoses;
* Age 12 years through 24 years, inclusive, at the time of consent;
* Engaged in care at the AMTU or its affiliate and/or partnering clinic. Individuals will be considered to be engaged in care if they have an AMTU (or its affiliate) clinic visit during the enrollment period;
* Ability to understand written and/or verbal English or Spanish.

Exclusion Criteria:

* Presence of serious psychiatric symptoms (e.g., active hallucinations, thought disorder) that would impair the individual's ability to complete the study measures;
* Visibly distraught (e.g., suicidal, homicidal, exhibiting violent behavior); or
* Intoxicated or under the influence of alcohol or other substances at the time of consent/assent

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All HIV-infected adolescents and young adults engaged in care at sites newly participating in ATN III and their affiliates who are between 12 and 24 years of age, inclusive, are aware of their HIV status and understand written and/or verbal English will be eligible for inclusion in the study. In addition, new patients who have their initial clinic visit within the enrollment period will also be eligible for participation
Sampling Method: Non-Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Collect information on for adolescents and young adults with HIV infection engaged in care at the AMTUs | 1 year
  Collect information on rates of adherence to medical regimens, sexual risk behavior, substance use and mental health concerns, along with basic demographic and biomedical data for adolescents and young adults with HIV infection engaged in care at the AMTUs to better understand the extent of risk behaviors as well as to understand risk and protective factors in this population.

SECONDARY OUTCOMES:
To better understand the complex relationships between adherence to medical regimens, sexual risk behavior, substance use and mental health concerns, and basic demographic and biomedical data in adolescents and young adults with HIV infection. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Heather Huszti, PhD, Study Chair — Adolescent Trials Network
Locations (5):
- United States (5):
  - University of Colorado Denver, Aurora, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - The Fenway Institute-Fenway Health, Boston, Massachusetts
  - Wayne State University-Children's Hospital of Michigan, Detroit, Michigan
  - Baylor College of Medicine - Pediatrics Allergy and Immunology, Houston, Texas

REFERENCES:
- See also: ATN Website — http://www.atnonline.org